CLINICAL TRIAL: NCT02964325
Title: Clinical Effectiveness of Conventional Versus Mirasol-treated Apheresis Platelets in Patients With Hypoproliferative Thrombocytopenia
Brief Title: Efficacy of Mirasol-treated Apheresis Platelets in Patients With Hypoproliferative Thrombocytopenia
Acronym: MIPLATE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Based interim analysis results, Data Monitoring Committee did not believe the primary efficacy endpoint would be met. No patient safety concerns.
Sponsor: Terumo BCTbio (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CTS-5030
Record Dates: First submitted 2016-11-09; First posted 2016-11-16 (Estimated); Results first posted 2021-07-16 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-07

CONDITIONS: Hematologic Malignancies; Hypoproliferative Thrombocytopenia
Keywords: hypoproliferative thrombocytopenia; hematologic malignancies; thrombocytopenia; platelet therapy; apheresis; pathogen reduction therapy
MeSH Terms: conditions — Hematologic Neoplasms; Thrombocytopenia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Though this is not a blinded study, treatment assignment is obtained through electronic system and should not be shared those performing the primary outcome assessment or assessors of adverse events.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Mirasol platelets (MIR PLTs) (Experimental): Leukoreduced, Trima Accel® apheresis platelets stored in 100% plasma, pathogen reduced with the Mirasol® Pathogen Reduction Technology (PRT) System
  Interventions: Device: Mirasol platelets (MIR PLTs)
- Reference platelets (REF PLTs) (Active Comparator): Leukoreduced, apheresis platelets stored in 100% plasma
  Interventions: Device: Reference platelets (REF PLTs)

INTERVENTIONS:
Device: Mirasol platelets (MIR PLTs) — The final product to be transfused to the subject will be leukoreduced (LR), apheresis (Aph) single-donor platelets (PLTs) at the standard therapeutic dose of 1 unit of Aph PLTs containing ≥ 3.0 × 1.0E11 PLTs. MIR PLTs will be treated with the Mirasol pathogen reduction technology system.
  Arms: Mirasol platelets (MIR PLTs)
Device: Reference platelets (REF PLTs) — The final product to be transfused to the subject will be LR-Aph single-donor PLTs at the standard therapeutic dose of 1 unit of Aph PLTs containing ≥ 3.0 × 1.0E11 PLTs.
  Arms: Reference platelets (REF PLTs)

SUMMARY:
This is a prospective, multi-center, controlled, randomized, non-inferiority study to evaluate the clinical effectiveness of Conventional versus Mirasol-treated apheresis platelets in subjects with hypoproliferative thrombocytopenia who are expected to have platelet count(s) ≤ 10,000/μL requiring ≥ 2 platelet transfusions.

DETAILED DESCRIPTION:
Patients will be randomized 1:1 to Mirasol-treated platelets (test platelets) or to conventional, untreated platelets (control platelets). The blood centers will collect the apheresis donor platelets and supply the test platelets to the hospital sites for transfusion into patients. Hospital sites will order control platelets as per their normal process, from their standard vendor.

The target population for the MIPLATE study are patients with hematologic malignancies with hypoproliferative thrombocytopenia who are expected to have platelet (PLT) count(s) of ≤ 10,000/μL requiring ≥ 2 PLT transfusions.

The primary objective of MIPLATE is to determine if the hemostatic efficacy of Mirasol-treated plasma stored Trima Accel® Aph PLTs are non-inferior to Conventional plasma stored Aph PLTs in subjects with hypoproliferative thrombocytopenia requiring PLT transfusions. The secondary objectives include comparing other efficacy and safety endpoints between the treatment groups.

Subjects with hematologic malignancies with hypoproliferative thrombocytopenia are anticipated to experience a "transfusion episode" where they will require PLT transfusion support until bone marrow recovery. During this period all PLT transfusions required for a study subject will be given according to the subject's treatment allocation for 28 days after the initial PLT transfusion OR until transfusion independence (10 days without PLT transfusion) prior to Day 28.

Additionally, serum samples for HLA antibody testing will be collected on Days 14, 28 and 56.

At a minimum, the initial post-randomization prophylactic PLT transfusion will be initiated for a PLT count ≤ 10,000/µL. Thereafter, indications for PLT transfusions may be PLT count-related prophylaxis, intervention-related prophylaxis, or therapeutic (treatment of active bleeding) as determined by the treating physician(s). The indication(s) for the transfusion(s) will be captured.

ELIGIBILITY:
Inclusion Criteria:

1. Weight > 10 kg (22 lbs)
2. Subject has a hematologic malignancy with hypoproliferative thrombocytopenia and is expected to have PLT count(s) ≤ 10,000/µL requiring ≥ 2 PLT transfusions
3. Laboratory results within 5 days prior to anticipated initiation of the first post randomization PLT transfusion:

   1. Prothrombin time (PT) and/or international normalized ratio (INR) ≤ 1.3 × the upper limit of normal (ULN)
   2. Activated partial thromboplastin time (aPTT) ≤ 1.3 × ULN
   3. Fibrinogen ≥ 100 mg/dL
4. Women of childbearing potential must have a negative pregnancy test and agree to practice a medically acceptable contraception regimen for the study duration. Women who are postmenopausal for at least 1 year (> 12 months since last menses) or are surgically sterilized do not require this test
5. IC from the subject or assent from the subject and consent from a parent or guardian, if the subject is < 18 years of age

Exclusion Criteria:

1. Treatment with pathogen-reduced blood products within previous 6 months
2. Subject has been previously enrolled in this study and received at least 1 per protocol PLT transfusion
3. a.) Subject is receiving therapeutic doses of antiplatelet agents, antifibrinolytics, and/or PLT specific growth factors within 10 days prior to randomization or b.) Subject is receiving therapeutic doses of anticoagulant, pro-coagulant or antithrombotic agents within 10 days prior to randomization. Subjects can be included if receiving the following: prophylactic dosing of anticoagulants (heparin, any low molecular weight heparin, enoxaparin, or fondaparinux), anticoagulants/thrombolytic agents used to maintain or re-establish the patency of catheters (heparin flushes or tissue-plasminogen activase [TPA], therapeutic doses of anticoagulants with a half-life of < 24 hours if it will be discontinued at least 24 hours prior to the first study transfusion, single periprocedural doses of anticoagulants with a half-life of < 24 hours or low dose aspirin (81 mg per day)
4. Subject has ≥ grade 2 bleeding at the time of randomization
5. Planned administration of bedside LR PLT transfusion(s)
6. Presently with or a history of acute promyelocytic leukemia (APML), idiopathic thrombocytopenic purpura (ITP), thrombotic thrombocytopenic purpura (TTP), or hemolytic uremic syndrome (HUS)
7. HLA and/or HPA-alloimmunization and/or platelet refractory as determined by the investigator
8. Hypersplenism as evidenced by splenomegaly based on investigator assessment at baseline
9. History or diagnosis of a disease affecting hemostasis
10. Currently taking, or participating in a clinical study involving PLT substitutes, PLT growth factors, or pharmacologic agents intended to enhance (i.e, antifibrinolytic agents) or decrease PLT hemostatic function
11. Acute or chronic medical disorder that, in the opinion of the investigator, would impair the ability of the subject to receive protocol treatment
12. Subject is pregnant or lactating
13. Inability of the subject to comply with study procedures and/or follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cortes, MD, Study Director — Terumo BCT; Sherrill Slichter, MD, Principal Investigator — Bloodworks Northwest
Locations (10):
- United States (10):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Health Shands Hospital, Gainesville, Florida
  - Emory University/Children's Hospital of Atlanta, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - John Hopkins University School of Medicine/Johns Hopkins Kimmel Cancer Center, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Robert Wood Johnson Medical School/RWJ University Hospital, New Brunswick, New Jersey
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred at 11 hospital sites within the US. Enrollment occurred between 05 MAY 2017 and 07 APR 2020.
Pre-assignment Details: Full Analysis Set (FAS) - all randomized subjects. Safety Set (SS) - randomized subjects who received at least 1 PLT transfusion post-randomization, independent of the outcome or successful completions of the procedure. Modified Intent-to-Treat (mITT) - all randomized subjects who had at least 1 study transfusion according to randomized study group. 422 subjects consented, 92 screen failed, 330 FAS, 28 received no transfusion, 302 SS, 5 received no transfusion per assigned group, 297 mITT.
Groups:
- MIRASOL: Randomized to leukoreduced, Trima Accel® apheresis platelets stored in 100% plasma, pathogen reduced with the Mirasol® Pathogen Reduction Technology (PRT) System
  Mirasol platelets (MIR PLTs): The final product to be transfused to the subject will be leukoreduced (LR), apheresis (Aph) single-donor platelets (PLTs) at the standard therapeutic dose of 1 unit of Aph PLTs containing ≥ 3.0 × 1.0E11 PLTs. MIR PLTs will be treated with the Mirasol pathogen reduction technology system.
- CONTROL: Randomized to leukoreduced, apheresis platelets stored in 100% plasma
  Reference platelets (REF PLTs): The final product to be transfused to the subject will be LR-Aph single-donor PLTs at the standard therapeutic dose of 1 unit of Aph PLTs containing ≥ 3.0 × 1.0E11 PLTs.
Period: Overall Study
Arm/Group | MIRASOL | CONTROL
Started | 164 | 166
Full Analysis Set (The Full Analysis Set (FAS) included all randomized subjects. Subjects were analyzed according to the treatment group to which they were assigned at randomization.) | 164 | 166
Modified Intent-to-Treat (The Modified Intent-to-Treat (mITT) Set included all randomized subjects who underwent at least 1 study transfusion post randomization according to the treatment group (MIRASOL or CONTROL) to which they were randomized.) | 145 | 152
Safety Set (The Safety Set (SS) included all randomized subjects who underwent at least 1 PLT transfusion post randomization, independent of the outcome or successful completion of the procedure. Subjects were analyzed according to the majority treatment (MIR PLTs or REF PLTs) received.) | 141 | 161
Completed | 143 | 143
Not Completed | 21 | 23
Not completed — Lost to Follow-up | 3 | 3
Not completed — Physician Decision | 5 | 4
Not completed — Death | 1 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Did not require PLT transfusion, had HLA positive | 10 | 12

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set was used for this analysis. Safety Set (SS) = randomized subjects who received at least 1 PLT transfusion post-randomization, independent of the outcome or successful completions of the procedure. Subjects were analyzed according to the majority treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | MIRASOL | CONTROL | Total
Number analyzed (Participants) | 141 | 161 | 302
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 10 | 16
  Between 18 and 65 years | 94 | 100 | 194
  >=65 years | 41 | 51 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (16.32) | 54.1 (18.24) | 54.4 (17.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 56 | 109
  Male | 88 | 105 | 193
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 130 | 147 | 277
  Unknown or Not Reported | 3 | 6 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Black or African American | 16 | 10 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 120 | 137 | 257
  Missing | 0 | 1 | 1
  Asian | 2 | 10 | 12
  Other | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 141 | 161 | 302
Height (cm) [Mean (Standard Deviation); unit: centimeters] | 170.29 (15.039) | 167.88 (18.472) | 169.01 (16.972)
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 86.96 (23.876) | 84.95 (25.400) | 85.89 (24.680)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: square meters] — The Dubois formula was used to calculate body surface area (BSA). BSA (m2) = 0.007184 × Height (cm)0.725 × Weight (kg)0.425
  square meters | 1.975 (0.3157) | 1.934 (0.3613) | 1.953 (0.3408)

OUTCOME MEASURES:

1. Primary Outcome: Days of ≥ Grade 2 Bleeding
Description: Number of days of Grade 2 or higher bleeding recorded from treatment start date through 28 days following the first transfusion, until transfusion independence (10 days without PLT transfusion) prior to Day 28, or study termination, whichever occurred first. Subjects who obtained transfusion independence prior to Day 28 were assumed to have zero bleeding events between the date of transfusion independence and Day 28. Observed and simulated data for off-protocol transfusion intervals were included.
Time Frame: From the first post-randomization platelet transfusion through 28 days following the first transfusion.
Population: The Modified Intent-to-Treat Analysis Set was used for this analysis. Modified Intent-to-Treat Analysis Set = all randomized subjects who had at least 1 study transfusion according to randomized study group.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MIRASOL | CONTROL
Number analyzed (Participants) | 145 | 152
Days | 1.7 (4.05) | 0.6 (1.51)
Statistical Analysis 1: Comparison: MIRASOL vs CONTROL; The MIRASOL and CONTROL groups were compared with respect to the number of days of WHO ≥ Grade 2 bleeding. This was carried out by fitting a negative binomial regression model with an offset defined as the natural logarithm (LN) of the number of days that bleeding was assessed in order to account for the fact that subjects had different numbers of bleeding assessment days; Test type: Non-Inferiority — An NI analysis was carried out to assess the primary efficacy endpoint with the null hypothesis being the MIRASOL group is inferior to the CONTROL group and the alternative hypothesis being the MIRASOL group is non-inferior to the CONTROL group. In this study, the NI margin was 1.6; Relative Rate = 2.79, 95% CI 2-sided [1.67 to 4.67] — The MIRASOL group represents the numerator and the CONTROL group represents the denominator for the relative rate. For days during off-protocol intervals, bleeding data were simulated using an estimate of the individual-specific bleeding rate

2. Secondary Outcome: Number and Percentage of Subjects With Human Leukocyte Antigen (HLA) Alloimmunization
Description: The outcome was the development of a new HLA Class I antibodies among subjects negative at baseline within each treatment group. Positivity for Class I HLA antibodies was determined by the 5 SD normalized background ratio cutoffs assay threshold (>59.2, LABScreen Mixed LSM12, One Lambda).
Time Frame: HLA antibodies were measured at Baseline and Days 14, 28, and 56.
Population: The Modified Intent-to-Treat Analysis Set was used for this analysis. Modified Intent-to-Treat Analysis Set = all randomized subjects who had at least 1 study transfusion according to randomized study group. Subjects who tested positive at the high assay threshold (5 SD normalized background ratio cutoffs >59.2, LABScreen Mixed LSM12, One Lambda) at Baseline were excluded from this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | MIRASOL | CONTROL
Number analyzed (Participants) | 136 | 141
Participants | 4 | 2

3. Secondary Outcome: Number and Percentage of Subjects With ≥ Grade 2 Bleeding
Description: The number and percentage of subjects with at least 1 day of ≥ Grade 2 bleeding from Day 0 through Day 27 (or until transfusion independence was achieved) by treatment group
Time Frame: From the first post-randomization platelet transfusion through 28 days following the first transfusion.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MIRASOL | CONTROL
Number analyzed (Participants) | 145 | 152
Participants | 58 | 46
Statistical Analysis 1: Comparison: MIRASOL vs CONTROL; The null hypothesis was H0: pt/pc > 1.2 (ie, MIRASOL had more than a 20% higher probability of a patient experiencing at least one WHO ≥ Grade 2 bleed compared to CONTROL); Test type: Non-Inferiority — A non-inferiority margin of 1.2 was used to evaluated this endpoint; p = 0.7274, Wald Non-inferiority Test; Relative Risk = 1.32, 95% CI 2-sided [0.97 to 1.81] — The MIRASOL group represents the numerator and the CONTROL group represents the denominator for the relative risk

4. Secondary Outcome: Number and Percentage of Subjects at the First Timepoint of ≥ Grade 2 Bleeding
Description: The time to first ≥ Grade 2 bleeding was analyzed using a log-rank test comparing survival curves stratified by treatment group.
Time Frame: From the first post-randomization platelet transfusion through 28 days following the first transfusion.
Population: The mITT Set was used for this analysis. Subjects that did not experience a ≥ Grade 2 bleed were censored at Day 27 or at date of transfusion independence (10th day without a PLT transfusion prior to last follow-up day or Day 27, whichever occurred earlier), where appropriate. Subjects that did not complete the study or were lost to follow-up were censored on the date of their last study visit in the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | MIRASOL | CONTROL
Number analyzed (Participants) | 145 | 152
Participants
  Day 4 | 115 | 128
  Day 8 | 92 | 110
  Day 12 | 72 | 85
  Day 16 | 33 | 48
  Day 20 | 11 | 27
  Day 24 | 5 | 13
  Day 28 | 4 | 11
Statistical Analysis 1: Comparison: MIRASOL vs CONTROL; Test type: Other; p = 0.07, Log-rank test

5. Secondary Outcome: Number and Percentage of Subjects With ≥ Grade 3 Bleeding
Description: The number and percentage of subjects with at least 1 day of ≥ Grade 3 bleeding from Day 0 through Day 27 (or until transfusion independence was achieved).
Time Frame: From the first post-randomization platelet transfusion through 28 days following the first transfusion.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MIRASOL | CONTROL
Number analyzed (Participants) | 145 | 152
Participants | 6 | 2
Statistical Analysis 1: Comparison: MIRASOL vs CONTROL; Test type: Other; p = 0.1649, Fisher Exact

6. Secondary Outcome: Number and Percentage of Subjects With PLT Refractoriness
Description: The number and percentage of subjects with PLT refractoriness defined as 2 sequential transfusions, each with corrected count increments (CCIs) < 5000 measured 1 hour post-transfusion.
Time Frame: From the first post-randomization platelet transfusion through 28 days following the first transfusion.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MIRASOL | CONTROL
Number analyzed (Participants) | 145 | 152
Participants | 41 | 20
Statistical Analysis 1: Comparison: MIRASOL vs CONTROL; Test type: Other; p = 0.0015, Fisher Exact; Risk Ratio (RR) = 2.15, 95% CI 2-sided [1.32 to 3.49]

7. Secondary Outcome: Number and Percentage of Subjects With Immune Platelet Refractoriness
Description: The number and percentage of subjects with PLT refractoriness for each treatment group. Subjects were defined as immune PLT refractoriness based on 2 sequential transfusion episodes, each with CCIs < 5000 measured 1 hour post transfusion, and who also had a positive antibody test within 14 days before or after the onset of PLT refractoriness.
Time Frame: Initial post-randomization platelet transfusion through high Class I HLA development.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MIRASOL | CONTROL
Number analyzed (Participants) | 136 | 141
Participants | 1 | 1

8. Other Pre Specified Outcome: Number and Percentage of Subjects With Unanticipated Adverse Device Effects (UADEs)
Description: UADEs are identified as treatment emergent adverse events reported by the investigator as serious, unanticipated, at least possibly related to study device or at least possibly related to treatment. UADEs were coded using Medical Dictionary for Regulatory Activities (MedDRA) Version 19.1
Time Frame: From initial post-randomization PLT transfusion through 72 hours following the last per protocol PLT transfusion.
Population: The Safety Set was used for this analysis. Safety Set = randomized subjects who received at least 1 PLT transfusion post-randomization, independent of the outcome or successful completions of the procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | MIRASOL | CONTROL
Number analyzed (Participants) | 141 | 161
Participants
  Blood and Lymphatic System Disorders/ Febrile Neutropenia | 1 | 0
  No UADEs | 140 | 161

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (SAEs) that occurred from initial post randomization platelet transfusion through seventy-two (72) hours following the transfusion end time of the last on-protocol PLT transfusion were reported. Deaths that occurred (including deaths due to bleeding) thirty days (30) following the transfusion end time of the last on-protocol PLT transfusion were reported.
Description: Treatment Emergent definition: an event that first appears during treatment, which was absent before or which worsened relative to the pre-treatment state. Treatment emergent are those events that occur during or following the first post-randomization PLT transfusion. All TEAEs/TESAEs were followed until resolution, stabilization, or the end of the subject's study participation which occurred first.
Arm/Group | MIRASOL | CONTROL
All-Cause Mortality (participants affected / at risk) | 1/141 | 3/161
Serious Adverse Events (participants affected / at risk) | 22/141 | 33/161
Other Adverse Events (participants affected / at risk) | 97/141 | 100/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MIRASOL (N=141) | CONTROL (N=161)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 11 (12)
Septic Shock (Infections and infestations) | 2 (2) | 2 (3)
Streptococcal bacteremia (Infections and infestations) | 2 (2) | 2 (2)
Bacteraemia (Infections and infestations) | 3 (3) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Stomatococcal infection (Infections and infestations) | 2 (2) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Cystitis viral (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Human herpesvirus 6 infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Septic arthritis staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Delayed engraftment (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transfusion-associated dyspnoea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transfusion-related circulatory overload (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transplant failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diaphragmatic hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0)
Engraftment syndrome (Immune system disorders) | 0 (0) | 1 (1)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Venoocclusive liver disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2) | 0 (0)
Blood culture positive (Investigations) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MIRASOL (N=141) | CONTROL (N=161)
Diarrhoea (Gastrointestinal disorders) | 21 (21) | 35 (35)
Vomiting (Gastrointestinal disorders) | 19 (19) | 14 (14)
Nausea (Gastrointestinal disorders) | 12 (12) | 8 (8)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 11 (11)
Stomatitis (Gastrointestinal disorders) | 11 (11) | 6 (6)
Pyrexia (General disorders) | 19 (20) | 16 (17)
Mucosal inflammation (General disorders) | 15 (15) | 19 (19)
Oedema peripheral (General disorders) | 15 (18) | 13 (14)
Fatigue (General disorders) | 13 (13) | 9 (9)
Febrile neutropenia (Blood and lymphatic system disorders) | 24 (27) | 17 (17)
Anaemia (Blood and lymphatic system disorders) | 12 (12) | 11 (11)
Hypokalaemia (Metabolism and nutrition disorders) | 14 (15) | 20 (20)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 8 (8)
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 (8) | 8 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 10 (10)
Headache (Nervous system disorders) | 9 (9) | 11 (12)
Dizziness (Nervous system disorders) | 7 (8) | 9 (11)
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 7 (13) | 8 (9)

LIMITATIONS AND CAVEATS:
The clinical trial was terminated early on the recommendation of the Data Monitoring Committee and in agreement with the Clinical Trial Steering Committee and the Sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/25/NCT02964325/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT02964325/SAP_001.pdf